CLINICAL TRIAL: NCT05879913
Title: Personalized Medical Treatment of Coronary Atherosclerosis in Prostate Cancer Patients Guided by Plaque Assessment With Quantitative Coronary CT Angiography (CCTA)
Brief Title: ASCVD Management Using CCTA in Prostate Cancer Patients on ADT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Comprehensive Cancer Network (Network); Pfizer (Industry); Sumitomo Pharmaceuticals America (Industry)
Responsible Party: Principal Investigator, Abhishek Khemka, Associate Professor of Clinical Medicine in Division of Cardiovascular Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTO-IUSCCC-0807
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Coronary Atherosclerosis; Quantitative Coronary CT Angiography; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CCTA Group (Experimental)
  Interventions: Device: Coronary CT Angiography (CCTA)
- Usual Care Group (No Intervention)

INTERVENTIONS:
Device: Coronary CT Angiography (CCTA) — Coronary computed tomographic angiography (CCTA) scan is a highly accurate noninvasive technique for detection of coronary artery plaque.
  Arms: CCTA Group

SUMMARY:
This is a randomized pilot study of Coronary CT Angiography (CCTA) for coronary atherosclerosis vs. Usual Care in patients with prostate cancer who are either planning to begin, or are currently taking androgen deprivation therapy (ADT) .

DETAILED DESCRIPTION:
This is a randomized pilot study where subjects are randomized 1:1 to either the CCTA group or non-CCTA (usual care) group. The target enrollment will be 100 subjects with accounting for a potential 10% dropout rate resulting in an sample size between 90-100 participants or 45-50per group arm.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information
2. Age ≥40 years at time of consent
3. Previous diagnosis of prostate cancer who are either currently receiving ADT, or who are planning to start ADT for >12 months
4. Patients currently on or planned for treatment with ADT plus androgen pathway inhibitor (abiraterone, enzalutamide, apalutamide, darolutamide) are allowed
5. ≥1 risk factor for ASCVD (hypertension, hyperlipidemia, diabetes, tobacco use)
6. No current cardiac symptoms

Exclusion Criteria:

1. Concurrent treatment with chemotherapy (docetaxel, cabazitaxel, mitoxantrone) at time of signing consent
2. Patient has implantable cardioverter-defibrillator (ICD), or pacemaker
3. History of coronary stents, obstructive coronary artery disease, myocardial infarction, coronary artery bypass grafting. History of atrial fibrillation
4. Renal dysfunction with creatinine clearance <35ml/min (calculated by Cockcroft-Gault Equation)
5. Allergy to iodinated contrast
6. Contraindication to the medications that may be given to regulate heart rate for the CCTA scan (applicable only to those randomized to the CCTA group)
7. Patients taking sildenafil or tadalafil for vasodilation, pulmonary hypertension, or BPH

   1. Note: Subjects taking sildenafil or tadalafil for erectile disfunction will still be eligible.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Atherosclerosis in CCTA Arm | Baseline
  Proportion of prostate cancer patients without cardiac symptoms in the CCTA arm who are reclassified into a higher risk group using automated plaque assessment from CCTA that would otherwise be classed as low risk for ASCVD using the PCE
Proportion of Subjects Eligible for Treatment Based on Automated Plaque Assessment from CCTA | Baseline
  Assessment of automated plaque from CCTA determining eligibility of lipid lowering treatment and aspirin

SECONDARY OUTCOMES:
Reduction in atherosclerotic cardiovascular disease (ASCVD) risk score | Baseline, 6 months, and 12 months
  Changes in risk over time with intensive medical treatment tailored to plaque burden to test results in a reduction in cardiovascular risk factors including blood pressure, glucose and lipid levels, thus reducing the ASCVD risk score.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Khemka, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana